CLINICAL TRIAL: NCT04257357
Title: Effect of an 8-week Supervised Exercise Programme on Physical Capacity and Quality of Life in Patients With Pulmonary Embolism. A Randomised Clinical Pilot Trial.
Brief Title: Supervised Exercise Following Pulmonary Embolism
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Covid-19 pandemia the study was never initiated
Sponsor: Central Jutland Regional Hospital (Other)
Collaborators: Aarhus University Hospital (Other); University of Aarhus (Other); VIA University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 6500012
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-02

CONDITIONS: Pulmonary Embolism
Keywords: Exercise; Quality of life; Physical capacity; Randomized trial; Pilot study
MeSH Terms: conditions — Pulmonary Embolism; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized clinical pilot trial with 8 weeks of follow-up
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Due to the intervention (exercise versus usual care) patients and trainers cannot be masked. Outcome assessors will be masked, as it will be different persons performing the 8-week follow-up, who have no knowledge of the group allocation. Furthermore, nurses and doctors providing usual care for the patients at the cardiologic departments are masked for group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Eight-week supervised exercise program: Patients in the intervention group receive the same usual care as the patients in the control group. In addition, the patients participate in an eight-week supervised interval training program. Briefly put, the patients are required to participate in at least 16 out of 20 possible training passes over the period of eight weeks. The training consists of a brief warm up followed by 35-50 minutes of interval training on a bicycle. The intensity and duration will increase over time
  Interventions: Behavioral: 8-weeks supervised exercise program
- Control group (Active Comparator): Patients in the control group receive usual care as a minimum. This includes three-five days of hospitalization where the anticoagulant treatment is initiated. The patient and the relatives receive general information about the disease and the course of treatment, the medication and future prevention of embolism. In the year following discharge the patient is booked for a check-up of their anticoagulant treatment with a physician or a nurse as required.
  It is considered an active comparator as all patients in the control group perform a watt-max cycle ergometer test with VO2 measurement 3 times, and this in it-self can influence patients' activity level.
  Interventions: Behavioral: Active control

INTERVENTIONS:
Behavioral: 8-weeks supervised exercise program — Please refer to group description
  Arms: Exercise group
Behavioral: Active control — Please refer to group description
  Arms: Control group

SUMMARY:
In a randomized controlled design the study aims to investigate whether an intervention of 8 weeks supervised bicycle training program in addition to usual care can positively influence the physical capacity and quality of life in patients medically treated for pulmonary embolism.

DETAILED DESCRIPTION:
Background:

The existing knowledge regarding pulmonary embolism is primarily focused on the diagnostic methods and medical treatment of the condition, and furthermore on the short term prognosis in terms of mortality and complications. Few studies have investigated the effect of exercise training on physical capacity and quality of life in patients struck by a pulmonary embolism, although many patients display worries and concerns about their physical and psychological wellbeing after discharge. Furthermore, a number of cross sectional studies and cohort studies have found some patients to have long-term reduced physical capacity and reduced quality of life following pulmonary embolism.

For the time being, no rehabilitation options are available for these patients neither in Denmark, or internationally. As no research exists regarding rehabilitation and exercise for these patients, the study will contribute with important knowledge in terms of what kind of exercise and physical tests we should provide in the future.

Methods and materials:

30 patients medically treated for pulmonary embolism will be recruited from three different hospitals. After inclusion and performance of baseline tests, the patients will be randomly allocated to either the control group, receiving standard care, or the intervention group, receiving an eight-week supervised interval training program in addition to standard care. At the time of inclusion and at the end of the training program (eight-weeks), the patient's physical capacity is measured using Vo2 Max test on an ergometer cycle and by the Incremental shuttle walk test. Furthermore, the patients complete a questionnaire on quality of life (Pulmonary Embolism Quality of Life Questionnaire and Euro-Qol 5 Dimensions), and also, daily physical activity during 7 days will be measured using accelerometry the week prior to baseline test, and the week following the 8-week test.

Statistical analysis:

For the primary outcome, change in physical capacity, parametrical statistics will be used to describe and analyse data (assuming these are normally distributed). For the secondary outcomes on quality oflife, these are ordinal scale data, and therefore will be described and analysed using non-parametrical statistics, while change in average physical activity level as measured with accelerometry and change in walking capacity as measured with the Incremental Shuttle Walk test will be measured using parametrical statistics, assuming a normal distribution of data.

As this is a pilot study the overall aim of the study is the estimate the potential effect of a supervise exercise program and further, to estimate the variance on the Watt-max test and VO2 max for this patient group, in order to calculate the needed sample size for a future full scale randomized controlled trial. In addition the aim of the pilot trial is to assess reach and feasibility of the intervention in this target group.

Expected outcomes and perspective:

The investigators expect that the supervised interval training program will increase the outcome of Vo2 Max, the incremental shuttle walk and PEQoL significantly compared to the control group receiving usual care. The feasibility of the intervention will be assessed, as well as recrution and retention rate of participants. The study will furthermore contribute significantly to the limited knowledge about the optimal rehabilitation for this group of patients and may thereby form the basis of future recommendations in this field.

ELIGIBILITY:
Inclusion Criteria:

1. Objective verified acute pulmonary embolism (ICD10 I260 and ICD10 I269), recurrent included.
2. Currently treated with anticoagulation medicine.
3. 18-80 years.
4. Speaking and understanding Danish.

Exclusion Criteria:

1. Pulmonary embolism found as a secondary finding scanning for other diseases.
2. In combination with severe comorbidity (e.g. cancer, COPD, heart disease, psychiatric disease like schizophrenia or bipolar disorder), pregnancy or being unable to complete Watt-max test and incremental shuttle walk test.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-20 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
VO2 max | Change from baseline test to 8 week follow-up (pre- to post-test)
  Change in physical capacity measured as VO2 max during watt-max test (cycle ergometer)

SECONDARY OUTCOMES:
Pulmonary Embolism Quality of Life | Change in score from baseline to 8 week follow-up
  The Pulmonary Embolism Quality of Life measures self-reported disease-related quality of life. The scale ranges from 0 (best) to 100 (worst).
EuroQol 5 Dimensions | Change in score from baseline to 8 week follow-up
  The EuroQol 5 Dimensions measures self-reported generic health-related quality of life. The 5-digit score is transformed to Time-Trade Off Values (TTO) using the Danish TTO-values, ranging from -0.64 (worst) to 1.000 (perfect health).
Incremental Shuttle-Walk Test | Change in number of meters walked from baseline to 8 week follow-up
  The Incremental Shuttle Walk test measures the number of meters walked on a 10 meter track. The walking speed is slow at the beginning of the test, and then eventually increases (using auditory beeps), reaching running speed at the end. The number of meters is counted, with 1200 meters being the maximum distance.
Average physical activity | Change in average daily physical activity (7 days) from baseline to 8 week follow-up
  The average daily activity level is measured as an average of 7 consecutive days using an accelerometer (a sensor), worn on the thigh. An average of 7 consecutive days prior to the baseline test and Again 7 consecutive days after the 8 week follow-up test

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Rolving, PhD, Study Chair — Central Jutland Hospital

IPD SHARING:
Plan to Share IPD: No
Due to the General Data Protection Regulations of EU we donot plan to make individual participant data available.